CLINICAL TRIAL: NCT03534804
Title: Cabozantinib Plus Pembrolizumab as First-Line Therapy for Cisplatin-Ineligible Advanced Urothelial Carcinoma (PemCab)
Brief Title: Cabozantinib Plus Pembrolizumab as First-Line Therapy for Cisplatin-Ineligible Advanced Urothelial Carcinoma
Acronym: PemCab
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: Exelixis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCI104688
Record Dates: First submitted 2018-05-11; First posted 2018-05-23 (Actual); Results first posted 2024-11-26 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Metastatic Urothelial Carcinoma; Bladder Cancer
MeSH Terms: conditions — Carcinoma, Transitional Cell; Urinary Bladder Neoplasms | interventions — cabozantinib; pembrolizumab

STUDY DESIGN:
Intervention Model Description: This is an open label, non-randomized phase 2 study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Cabozantinib and Pembrolizumab, all patients (Experimental)
  Interventions: Drug: Cabozantinib; Drug: Pembrolizumab

INTERVENTIONS:
Drug: Cabozantinib — Cabozantinib is administered at 40 mg oral daily
  Other Names: XL184
Drug: Pembrolizumab — Pembrolizumab will be administered at a fixed dose of 200mg intravenously every 3 weeks.

SUMMARY:
This is an open label, non-randomized phase 2 study of the combination of pembrolizumab and cabozantinib to assess overall response rate (ORR), progression free survival at 6 months (PFS6), and overall survival (OS) in patients with metastatic urothelial carcinoma (UC) ineligible for cisplatin.

ELIGIBILITY:
Pre-Screening Eligibility

* Male or female subject aged ≥ 18 years.
* Clinically, subject is a candidate for urothelial diagnostic procedure (fresh soft-tissue biopsy or TURBT).
* Subject meets general medical criteria for consideration of treatment with immunotherapy using a checkpoint inhibitor.

Treatment Inclusion Criteria:

* Histologically proven transitional cell or urothelial carcinoma.
* Patients with locally advanced or metastatic urothelial carcinoma must meet one of the following:

  * Patients who are not eligible for cisplatin-containing chemotherapy AND whose tumors express PD-L1 (Combined Positive Score (CPS) ≥ 10 as determined by an FDA-approved test; OR
  * Patients who are not eligible for any platinum-containing chemotherapy regardless of PD-L1 status.
* Metastatic (any N+ or M1) or locally advanced, unresectable (T4bN0) disease.
* Measurable disease is required as determined by RECIST v1.1.
* Performance Status ECOG 0-2
* Cisplatin-ineligibility based on ≥1 of the following:

  * Estimated creatinine clearance between ≥30 and <60 ml/min (Cockcroft-Gault formula)
  * ECOG PS>1
  * Hearing loss
  * Baseline neuropathy > grade 1.
  * Patient refusal
* Be greater to or equal to 18 years of age on day of signing informed consent.
* Serum albumin ≥ 2.8 g/dl
* Alkaline phosphatase (ALP) ≤ 3 × upper limit of normal (ULN). ALP ≤ 5 × ULN with documented bone metastases.
* Negative serum or urine pregnancy test at screening for women of childbearing potential.
* Highly effective contraception for both male and female subjects throughout the study and for at least 120 days after last pembrolizumab treatment administration if the risk of conception exists.
* Must have recovered from adverse effects of any prior surgery, radiotherapy or other antineoplastic therapy to grade ≤ 2. If notrecovered to grade ≤ 2, these must be deemed to be irreversible adverse events related to prior surgery and/or radiation therapy (such as incontinence or sexual dysfunction) per investigator clinical judgment.
* Recovery to baseline or ≤ Grade 2 CTCAE v5 from toxicities related to any prior treatments, unless AE(s) are clinically nonsignificant and/or stable on supportive therapy. Alopecia, sensory neuropathy Grade ≤ 2, or other Grade ≤ 2 not constituting a safety risk based on investigator's judgment are acceptable.
* Last dose of any radiation therapy > 2 weeks before first dose of study treatment.
* Able to provide informed consent and willing to sign an approved consent form that conforms to federal and institutional guidelines.
* Adequate organ function as defined in the protocol

Exclusion Criteria:

* Prior chemotherapy for metastatic urothelial carcinoma.
* Prior chemotherapy for localized urothelial carcinoma that has been completed less than 6 months before registration.
* Variant histologies other than urothelial carcinoma will not be allowed. Patients with a component of variant histologies will be allowed to enroll, if urothelial carcinoma is the predominant histology per investigator judgement. Patients with any component of small cell will be excluded.
* Has received prior treatment with cabozantinib.
* Receipt of any type of small molecule kinase inhibitor (including investigational kinase inhibitor) within 2 weeks before first dose of study treatment.
* Receipt of any type of cytotoxic, biologic, or other systemic anticancer therapy (including investigational) within 4 weeks before first dose of study treatment.
* Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent or other checkpoint inhibitors previously.
* Radiation therapy for bone metastasis ≤ 2 weeks, any other radiation therapy within 4 weeks before first dose of study treatment. Systemic treatment with radionuclides within 6 weeks before the first dose of study treatment. Subjects with clinically relevant ongoing complications from prior radiation therapy are not eligible.
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least 4 weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability.
* Concomitant anticoagulation with oral anticoagulants except for those specified below.

Allowed anticoagulants are the following:

* Prophylactic use of low-dose aspirin for cardioprotection (per local applicable guidelines) is permitted.
* Low-dose low molecular weight heparins (LMWH) are permitted.
* Therapeutic doses of LMWH or anticoagulation with direct factor Xa inhibitors rivaroxaban, edoxaban, or apixaban is allowed in subjects without known brain metastases who are on a stable dose of the anticoagulant for at least 1 week before the first dose of study treatment without, clinically significant hemorrhagic complications from the anticoagulation regimen or the tumor.

  * The subject has prothrombin time (PT)/INR or partial thromboplastin time (PTT) test ≥ 1.3 × ULN within 14 days before the first dose of study treatment.
  * The subject has uncontrolled, significant intercurrent or recent illness including, but not limited to, the following conditions:
* Cardiovascular disorders:

  * Ongoing congestive heart failure exacerbation or New York Heart Association Class 4, unstable angina pectoris, serious cardiac arrhythmias.
  * Uncontrolled hypertension defined as sustained blood pressure (BP) > 150 mm Hg systolic or > 100 mm Hg diastolic despite optimal antihypertensive treatment. Uncontrolled hypertension needs to be determined based on persistently high blood pressure readings over more than 24 hours and should NOT be based on the blood pressure readings from one clinic visit. Blood pressure readings done at home or by primary care providers are acceptable. If a blood pressure reading on the day of screening is high, but there are documented acceptable ( ≤150 mm Hg systolic and ≤100 mm Hg diastolic) blood pressure readings prior to or after the screening visit (with or without the use of anti-hypertensive medications), patient will not be considered to have uncontrolled hypertension.
  * Stroke (including transient ischemic attack [TIA]), myocardial infarction (MI), or other ischemic event, or symptomatic thromboembolic event (eg, deep venous thrombosis, pulmonary embolism) occurring less than or equal to 6 months before first dose of cabozantinib. [Note: Subjects with a diagnosis of deep vein thrombosis (DVT) or incidentally detected asympotmatic and sub-segmental pulmonary embolism (PE) on routine scans are allowed if on a stable dose of anti-coagulation for at least 1 week before first dose of study treatment].

    * Clinically significant hematuria, hematemesis, or hemoptysis of > 0.5 teaspoon (2.5 ml) of red blood, or other history of significant bleeding (eg, pulmonary hemorrhage) within 12 weeks before first dose.
* Gastrointestinal (GI) disorders including those associated with a high risk of perforation or fistula formation:

  * The subject has evidence of tumor invading the GI tract, active peptic ulcer disease, inflammatory bowel disease (eg, Crohn's disease), diverticulitis, cholecystitis, symptomatic cholangitis or appendicitis, acute pancreatitis, acute obstruction of the pancreatic duct or common bile duct, or gastric outlet obstruction.
  * Abdominal fistula, GI perforation, bowel obstruction, or intra-abdominal abscess within 6 months before first dose.

Note: Complete healing of an intra-abdominal abscess must be confirmed before first dose.

* Cavitating pulmonary lesion(s) or known endotracheal or endobronchial disease manifestation.
* Lesions invading or encasing any major blood vessels.
* Other clinically significant disorders that would preclude safe study participation per investigator clinical judgement.

  * Serious non-healing wound/ulcer/bone fracture.
  * Uncompensated/symptomatic hypothyroidism.
  * Moderate to severe hepatic impairment (Child-Pugh B or C).

    * Other severe acute or chronic medical conditions including immune colitis, inflammatory bowel disease, immune pneumonitis, pulmonary fibrosis or psychiatric conditions including recent (within the past year) or active suicidal ideation or behavior; or laboratory abnormalities that may increase the risk associated with study participation or study treatment administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the patient inappropriate for entry into this study.
    * Major surgery (eg, GI surgery, removal or biopsy of brain metastasis) within 8 weeks before first dose of study treatment. Complete wound healing from major surgery must have occurred 1 month before first dose and from minor surgery (eg, simple excision, tooth extraction) at least 10 days before first dose. Subjects with clinically relevant ongoing complications per investigator clinical judgement from prior surgery are not eligible.
    * Corrected QT interval calculated by the Fridericia formula (QTcF) > 500 ms per electrocardiogram (ECG) within 28 days before first dose of study treatment.

Note: If a single ECG shows a QTcF with an absolute value > 500 ms, two additional ECGs at intervals of approximately 3 min must be performed after the initial ECG, and the average of these three consecutive results for QTcF will be used to determine eligibility.

* Diagnosis of another malignancy within 2 years before first dose of study treatment, with the exception of those determined by the treating investigator to have a negligible risk of metastasis or death (such as adequately treated carcinoma in situ of the cervix, basal or squamous cell skin cancer, ductal carcinoma in situ treated surgically with curative intent, localized prostate cancer treated with curative intent and/or no intent for further treatment, or incidental prostate cancer)
* Current use of immunosuppressive medication, EXCEPT for the following: a. intranasal, inhaled, topical steroids, or local steroid injection (e.g., intra-articular injection); b. Systemic corticosteroids at physiologic doses ≤ 10 mg/day of prednisone or equivalent; c. Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication).
* Has active autoimmune disease currently requiring systemic treatment with high dose corticosteroids (dose more than physiologic replacement doses equivalent to prednisone 10 mg daily) or (disease modifying immunosuppressive agents). Replacement therapy (e.g. thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, intranasal, inhaled, topical steroids, or local steroid injection) is not considered an exclusion.
* Active autoimmune disease that might deteriorate significantly when receiving an immuno-stimulatory agent per treating physician's clinical judgment. Subjects with diabetes type I, vitiligo, psoriasis, or hypo- or hyperthyroid diseases not requiring immunosuppressive treatment are eligible.
* Prior organ transplantation including allogenic stem-cell transplantation.
* Has known history of (non-infectious) pneumonitis that required steroids or has current pneumonitis.
* Has an active infection currently requiring systemic (intravenous) antibiotic therapy.
* Has a known history of active TB (Bacillus Tuberculosis).
* Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
* Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
* Active and inactive vaccinations within 4 weeks of the first dose of pembrolizumab is prohibited.
* Known prior severe hypersensitivity to investigational products or any component in its formulations, including known severe hypersensitivity reactions to monoclonal antibodies (NCI CTCAE v4.03 Grade ≥ 3).
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
* Subjects taking prohibited medications as described in Section 6.8. A washout period of prohibited medications for a period of at least two weeks or as clinically indicated should occur prior to the start of treatment.
* Inability to swallow tablets or evidence of impaired intestinal absorption Previous systemic chemotherapy treatment for urothelial carcinoma, with the exception of perioperative chemotherapy treatment alone or with concurrent radiation within 6 months prior to treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2018-09-18 (Actual); Primary Completion 2023-08-02 (Actual); Study Completion 2024-04-15 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Moffitt Cancer Center, Tampa, Florida
  - Winship Cancer Institute, Emory University, Atlanta, Georgia
  - Huntsman Cancer Institute, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 36 participants received study treatment. Adverse event collection started at consent, hence there is additional one participant who experienced an SAE during screening and did not enroll in the study.
Groups:
- Cabozantinib and Pembrolizumab, All Patients: Cabozantinib: Cabozantinib was administered at 40 mg oral daily.
  Pembrolizumab: Pembrolizumab was administered at a fixed dose of 200mg intravenously every 3 weeks.
Period: Overall Study
Arm/Group | Cabozantinib and Pembrolizumab, All Patients
Started | 36
Completed | 35
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Cabozantinib and Pembrolizumab, All Patients
Number analyzed (Participants) | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.06 (7.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 32
  Unknown or Not Reported | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 34
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 36
ECOG at Baseline [Count of Participants; unit: Participants]
  Fully Active | 11
  Restricted | 21
  Ambulatory | 4
  Capable of limited selfcare | 0
  Completely disabled | 0
  Dead | 0
  Not Done | 0
Overall Stage at Enrollment [Count of Participants; unit: Participants] — Staging systems are utilized in cancer care to standardize the extent of the cancer. The TNM (Tumor, Nodes, Metastasized) system is used for bladder cancer. With this system, the overall stage is numbered from 0 to 4.
  Stage 1 means cancer has not spread to the muscle (Tis+N0+M0).
  Stage 2 means the cancer has spread to the muscle (T1+N0+M0).
  Stage 3 means cancer has spread through the bladder to nearby tissues (T3+N0+M0).
  Stage 4 is cancer which has spread to distant lymph nodes or organs (T4+NX+M0), (T4+N0+M0), (Any T+N1+M0), (Any T+N2+M0), or (Any T+Any N+M1).
  Participants
    I: cancer has not spread to the muscle (Tis+N0+M0). | 1
    III: cancer has spread through the bladder to nearby tissues (T3+N0+M0) | 1
    IIIA: cancer has spread to the fat surrounding the bladder (T3a/T3b/T4a+N0+M0) or (T1-4a, N1+M0). | 1
    IV: cancer spread to far lymph nodes or organs (T4+NX/N0+M0), (Any T+N1/N2+M0), or (Any T+Any N+M1). | 27
    IVA: cancer spread to the pelvic or abdominal wall (T4b + Any N + M0) or (Any T + Any N + M1a). | 1
    IVB: cancer spread to distant organs (Any T + Any N + M1b) | 2
    Unknown/Unable to Determine | 3
Primary Location of Disease [Count of Participants; unit: Participants]
  Lower Tract | 17
  Upper Tract | 18
  Upper and Lower Tract | 1
Height [Mean (Standard Deviation); unit: cm] | 173.66 (9.84)
Weight [Mean (Standard Deviation); unit: kg] | 90.36 (26.74)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 29.71 (7.44)
Smoking Status [Count of Participants; unit: Participants]
  Current Smoker | 4
  Former Smoker | 19
  Non-Smoker | 13
History of Hypertension [Count of Participants; unit: Participants]
  No | 7
  Yes | 29
T Stage at Enrollment [Count of Participants; unit: Participants] — Staging systems are utilized in cancer care to standardize the extent of the cancer. The TNM (Tumor, Nodes, Metastasized) system is used for bladder cancer. With this system, T describes how far the primary tumor has grown and if it has grown into nearby tissue. This staging system ranges from T0 (No evidence of a primary tumor) to T4 (The tumor has grown outside the bladder to other organs).
  Participants
    T0: There is no evidence of a primary tumor. | 3
    T1: The cancer has grown into the connective tissue of the bladder but not the muscle layer. | 8
    T1a: A subset of T1 in which the tumor has not grown into the muscular mucosae-vascular plexus. | 1
    T2: The cancer has grown into the bladder's muscle layer, but it has not reached fatty tissue layer. | 6
    T3: The cancer grew into the bladder's fatty tissue layer but not into the pelvic or abdominal wall. | 5
    T4: The cancer has grown through the bladder into the pelvic or abdominal wall. | 4
    Tx: Insufficient information to assess the tumor. | 8
    Unknown/Unable to Determine | 1
N Stage at Enrollment [Count of Participants; unit: Participants] — Staging systems are utilized in cancer care to standardize the extent of the cancer. The TNM (Tumor, Nodes, Metastasized) system is used for bladder cancer. With this system, N describes if any cancer spread to lymph nodes.
  This staging system ranges from N0 (no regional lymph node spread) to N3 (cancer cells have spread to one or more lymph node).
  Participants
    N0: The cancer did not spread to lymph nodes. | 13
    N1: The cancer spread to 1 lymph node in the pelvis. | 5
    N2: The cancer spread to 2 or more lymph nodes in the pelvis. | 5
    N3: The cancer spread to lymph nodes farther away from the bladder (along the common iliac arteries) | 4
    NX: Due to lack of information, regional lymph nodes could not be assessed. | 7
    Unknown/Unable to Determine | 2
M Stage at Enrollment [Count of Participants; unit: Participants] — Staging systems are utilized in cancer care to standardize the extent of the cancer. The TNM (Tumor, Nodes, Metastasized) system is used for bladder cancer. With this system, M describes if any cancer spread to other parts of the body.
  This staging system ranges from M0 (the cancer has not spread to other parts of the body) to M1b (the cancer has spread to one or more distant organs like the bones, liver, or lungs).
  Participants
    M0: The cancer has not spread to other parts of the body. | 4
    M1: The cancer has spread to other parts of the body. | 21
    M1a: The cancer has spread to distant lymph nodes. | 2
    M1b: The cancer has spread to 1 or more distant organs. | 3
    MX: Due to a lack of information, metastasis could not be assessed. | 3
    Unknown/Unable to Determine | 3
Histology [Count of Participants; unit: Participants]
  Mixed | 8
  Pure Urothelial | 28
Prior Chemotherapy [Count of Participants; unit: Participants]
  Yes | 10
  No | 26
Prior Bacillus Calmette-Guerin (BCG) Treatment [Count of Participants; unit: Participants]
  Yes | 10
  No | 26

OUTCOME MEASURES:

1. Primary Outcome: Count of Participants With Response Measured by RECIST 1.1
Description: To evaluate measurable disease overall response. Subjects were evaluated by CT scans at regular intervals for disease assessment by RECISTv1.1 criteria for the duration of treatment.
  Response Evaluation Criteria in Solid Tumors (RECIST) is a standard measure of how well cancer patients respond to treatment. Possible scores are CR (Complete Response; total disappearance of all target lesions), PR (Partial Response; at least a 30% decrease of the sum of the longest diameter of all target lesions), PD (Progressive Disease; at least a 20% increase of the sum of the longest diameter of all target lesions), and SD (Stable Disease; neither a sufficient decrease for PR, or sufficient increase for PD). Overall response is the count of PR and CR scores among the participants' best RECISTv1.1 responses.
Time Frame: From baseline disease assessment to best response disease assessment, measured up to 28 months.
Population: Of the 36 participants enrolled in the trial, one participant withdrew prior to reaching this endpoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Cabozantinib and Pembrolizumab, All Patients
Number analyzed (Participants) | 35
Participants | 16

2. Secondary Outcome: Count of Participants Who Were Progression-free at the Completion of Study Follow-up (PFS).
Description: To evaluate progression-free survival at completion of study follow-up (PFS). PFS is defined as the count of participants who remained alive and progression-free completion of their follow-up period. Participants were followed up to six months after completion of the study treatment.
  Subjects were evaluated by CT scans at regular intervals for disease assessment by RECISTv1.1 criteria (as described in the primary outcome) for the duration of treatment.
Time Frame: Up to 34 months from the start of the study treatment.
Population: Of the 36 participants enrolled in the trial, one participant withdrew prior to reaching this endpoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Cabozantinib and Pembrolizumab, All Patients
Number analyzed (Participants) | 35
Participants | 18

3. Secondary Outcome: Count of Overall Survival (OS) at Completion of Study Follow-up
Description: To evaluate Overall Survival (OS) at completion of study follow-up. OS is defined as the count of participants who remained alive after their follow-up period. Participants were followed up to six months after completion of the study treatment.
  Subjects were followed via telephone contact or medical record review for survival 6 months after completing the study treatment.
Time Frame: Up to 34 months from the start of the study treatment.
Population: Of the 36 participants enrolled in the trial, one participant was not evaluable for efficacy endpoints.
Measure: Count of Participants; unit: Participants
Arm/Group | Cabozantinib and Pembrolizumab, All Patients
Number analyzed (Participants) | 35
Participants | 23

4. Secondary Outcome: Occurrence of Adverse Events and Serious Adverse Events
Description: To evaluate toxicities associated with the combination treatment. Subjects were monitored for adverse events from the start of treatment through 30 days after the last dose of study treatment, and serious adverse events were collected until 90 days after the cessation of study treatment.
  The severity of adverse events was assessed using CTCAE v5.0 criteria, a 1-5 scale with higher numbers indicating greater severity. Grade 1 indicates "mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated" and Grade 5 indicates "death related to AE". The treating investigator evaluated each adverse event to assess its attribution to the study treatment.
  This outcome measure will report the following:
  * The count of participants who had a grade 1-2 event, related to study treatment.
  * The count of the participants who had a grade 3-4 event, related to study treatment.
  * The count of the participants who had a grade 5 event or higher,
Time Frame: Up to 31 months from the start of study treatment.
Population: All participants who received the study drug were evaluated for adverse events and serious adverse events endpoints.
Measure: Count of Participants; unit: Participants
Arm/Group | Cabozantinib and Pembrolizumab, All Patients
Number analyzed (Participants) | 36
Participants
  Count of participants with a related grade 1-2 event. | 23
  Count of participants with a related grade 3-4 event. | 6
  Count of participants with a related grade 5 event or higher. | 0

ADVERSE EVENTS:
Time Frame: Collection of Non-Serious Adverse Events (NSAE) began after informed consent and ended 30 days post the last dose of study treatment. Collection of Serious Adverse Events (SAE) began after informed consent and ended 90 days after the last dose of study treatment or until new cancer treatment was initiated. Patients were followed for survival 6 months after study treatment. NSAEs were assessed up to 29 months, SAEs up to 31 months, and death up to 34 months from the start of treatment.
Description: Information about all adverse events, whether volunteered by the subject, discovered by investigator questioning, or detected through physical examination, laboratory test or other means, was collected and recorded at every study visit.
Arm/Group | Cabozantinib and Pembrolizumab, All Patients
All-Cause Mortality (participants affected / at risk) | 12/37
Serious Adverse Events (participants affected / at risk) | 22/37
Other Adverse Events (participants affected / at risk) | 37/37
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cabozantinib and Pembrolizumab, All Patients (N=37)
Acute kidney injury (Renal and urinary disorders) | 2 (2)
Alanine aminotransferase increased (Investigations) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Atrial flutter (Cardiac disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (2)
Bladder perforation (Renal and urinary disorders) | 1 (3)
Cardiac disorders - Other, specify (Cardiac disorders) | 1 (1) — bradycardia
Chest pain - cardiac (Cardiac disorders) | 1 (1)
Colonic perforation (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Disease progression (General disorders) | 2 (2)
Encephalopathy (Nervous system disorders) | 1 (1)
Guillain-Barre syndrome (Nervous system disorders) | 1 (1)
Heart failure (Cardiac disorders) | 1 (1)
Hematuria (Renal and urinary disorders) | 3 (3)
Hepatitis viral (Infections and infestations) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Immune system disorders - Other, specify (Immune system disorders) | 1 (1) — Immune-mediated hepatitis
Infections and infestations - Other, specify (Infections and infestations) | 1 (1) — Left psoas abscess
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1 (1) — Chronic pain
Paroxysmal atrial tachycardia (Cardiac disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Rectal hemorrhage (Gastrointestinal disorders) | 1 (1)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1 (1) — Urinary tract obstruction
Sepsis (Infections and infestations) | 1 (1)
Thromboembolic event (Vascular disorders) | 6 (6)
Urinary tract infection (Infections and infestations) | 3 (4)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cabozantinib and Pembrolizumab, All Patients (N=37)
Abdominal distension (Gastrointestinal disorders) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 4 (5)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1)
Agitation (Psychiatric disorders) | 1 (1)
Alanine aminotransferase increased (Investigations) | 4 (12)
Alkaline phosphatase increased (Investigations) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2)
Anemia (Blood and lymphatic system disorders) | 7 (10)
Anorexia (Metabolism and nutrition disorders) | 13 (16)
Anosmia (Nervous system disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (9)
Aspartate aminotransferase increased (Investigations) | 5 (12)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Bladder spasm (Renal and urinary disorders) | 2 (2)
Bloating (Gastrointestinal disorders) | 3 (3)
Blood bilirubin increased (Investigations) | 1 (2)
Blood lactate dehydrogenase increased (Investigations) | 1 (1)
Blurred vision (Eye disorders) | 3 (4)
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 1 (1)
Cardiac disorders - Other, specify (Cardiac disorders) | 1 (1)
Cardiac troponin I increased (Investigations) | 2 (2)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Chills (General disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Cognitive disturbance (Nervous system disorders) | 1 (2)
Colitis (Gastrointestinal disorders) | 1 (1)
Concentration impairment (Nervous system disorders) | 1 (1)
Confusion (Psychiatric disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 15 (17)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Creatinine increased (Investigations) | 2 (3)
Depression (Psychiatric disorders) | 1 (2)
Diarrhea (Gastrointestinal disorders) | 24 (42)
Dizziness (Nervous system disorders) | 3 (4)
Dry eye (Eye disorders) | 1 (1)
Dry mouth (Gastrointestinal disorders) | 4 (4)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 8 (9)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 9 (10)
Dysuria (Renal and urinary disorders) | 2 (2)
Ear and labyrinth disorders - Other, specify (Ear and labyrinth disorders) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 1 (1)
Edema limbs (General disorders) | 3 (4)
Electrocardiogram QT corrected interval prolonged (Investigations) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1)
Endocrine disorders - Other, specify (Endocrine disorders) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Eye disorders - Other, specify (Eye disorders) | 1 (1)
Eye pain (Eye disorders) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 2 (2)
Fatigue (General disorders) | 23 (38)
Fecal incontinence (Gastrointestinal disorders) | 1 (1)
Fever (General disorders) | 2 (2)
Flank pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Flatulence (Gastrointestinal disorders) | 2 (2)
Flu like symptoms (General disorders) | 1 (1)
Gait disturbance (General disorders) | 1 (1)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2 (2)
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 4 (4)
General disorders and administration site conditions - Other, specify (General disorders) | 1 (1)
Generalized edema (General disorders) | 2 (2)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 3 (5)
Hair color changes (Skin and subcutaneous tissue disorders) | 3 (3)
Headache (Nervous system disorders) | 6 (6)
Hematuria (Renal and urinary disorders) | 5 (10)
Hemorrhoids (Gastrointestinal disorders) | 3 (3)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 10 (12)
Hypercalcemia (Metabolism and nutrition disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 (2)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 1 (2)
Hyperparathyroidism (Endocrine disorders) | 1 (1)
Hypertension (Vascular disorders) | 5 (8)
Hyperthyroidism (Endocrine disorders) | 2 (3)
Hypocalcemia (Metabolism and nutrition disorders) | 3 (5)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalemia (Metabolism and nutrition disorders) | 3 (5)
Hypomagnesemia (Metabolism and nutrition disorders) | 9 (11)
Hyponatremia (Metabolism and nutrition disorders) | 2 (8)
Hypophosphatemia (Metabolism and nutrition disorders) | 10 (24)
Hypotension (Vascular disorders) | 2 (2)
Hypothyroidism (Endocrine disorders) | 9 (11)
Immune system disorders - Other, specify (Immune system disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 5 (6)
Investigations - Other, specify (Investigations) | 11 (15)
Lethargy (Nervous system disorders) | 1 (1)
Lipase increased (Investigations) | 1 (1)
Lung infection (Infections and infestations) | 1 (1)
Malaise (General disorders) | 1 (1)
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 9 (12)
Muscle cramp (Musculoskeletal and connective tissue disorders) | 4 (4)
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 19 (26)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Oral dysesthesia (Gastrointestinal disorders) | 7 (8)
Oral pain (Gastrointestinal disorders) | 1 (1)
Pain (General disorders) | 6 (8)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3)
Palmar-plantar erythrodysesthesia syndrome (Skin and subcutaneous tissue disorders) | 14 (25)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Paresthesia (Nervous system disorders) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (2)
Platelet count decreased (Investigations) | 2 (4)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (3)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (4)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Proteinuria (Renal and urinary disorders) | 5 (13)
Pruritus (Skin and subcutaneous tissue disorders) | 13 (15)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 (4)
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 5 (7)
Reproductive system and breast disorders - Other, specify (Reproductive system and breast disorders) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1 (4)
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1)
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 6 (11)
Skin atrophy (Skin and subcutaneous tissue disorders) | 1 (1)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1)
Stomach pain (Gastrointestinal disorders) | 1 (1)
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 2 (2)
Syncope (Nervous system disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1)
Thrush (Infections and infestations) | 1 (1)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Upper respiratory infection (Infections and infestations) | 2 (2)
Urinary frequency (Renal and urinary disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (2)
Urinary tract infection (Infections and infestations) | 10 (15)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1)
Urine output decreased (Investigations) | 1 (1)
Vascular disorders - Other, specify (Vascular disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 11 (13)
Weight loss (Investigations) | 8 (12)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Agreement with UNIVERSITY OF UTAH and MOFFITT CANCER CENTER:

University and PI shall have first right to publish and disseminate the results of their investigative findings under the Study unless 18 months have elapsed following completion of the Study without such publication by University or PI.

Agreement with UNIVERSITY OF UTAH and EMORY UNIVERSITY:

University and PI shall have first right to publish and disseminate the results of their investigative findings under the Study.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-30): https://cdn.clinicaltrials.gov/large-docs/04/NCT03534804/Prot_SAP_000.pdf